CLINICAL TRIAL: NCT02505334
Title: A Trial Comparing the Efficacy and Safety of Liraglutide 1.8 mg/Day to Liraglutide 0.9 mg/Day in Japanese Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-4174; U1111-1164-5462 (Other: WHO); JapicCTI-152975 (Registry Identifier: JAPIC)
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liraglutide 1.8 mg (Experimental): The total trial duration for the 1.8 mg/day treatment arm will be approximately 67 weeks, consisting of 2 weeks screening period, a 12 weeks run-in period, a 26-week main treatment period, a safety extension period of 26 weeks and a follow-up visit.
  Interventions: Drug: liraglutide
- Liraglutide 0.9 mg (Active Comparator): The total trial duration for the 0.9 mg/day treatment arm will be approximately 41 weeks, consisting of 2 weeks screening period, a 12 weeks run-in period, a 26-week treatment period, and a follow-up visit.
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Injected subcutaneously s.c. (under the skin) once daily.

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to compare the efficacy and safety of liraglutide 1.8 mg/day to liraglutide 0.9 mg/day in Japanese subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese subjects at least 20 years of age at the time of informed consent
* Type 2 diabetes subjects (diagnosed clinically) for at least 6 months prior to screening
* HbA1c 7.5-10.0% [58 mmol/mol-86 mmol/mol] (both inclusive)
* Subjects on stable therapy with one OAD (oral antidiabetic drug) (stable therapy is defined as unchanged medication and unchanged dose) for for at least 60 days before screening according to approved Japanese labelling

Exclusion Criteria:

* Treatment with insulin within 12 weeks prior to screening
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 60 days before screening
* Screening calcitonin equal or above 50 ng/l
* History of pancreatitis (acute or chronic)
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN 2)
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV
* Within the past 180 days any of the following: myocardial infarction, stroke or hospitalisation for unstable angina and/or transient ischemic attack
* Diagnosis of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer, polyps and in-situ carcinomas)
* Any condition which, in the opinion of the investigator might jeopardise subject's safety or compliance with the protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (37):
- Japan (37):
  - Novo Nordisk Investigational Site, Annaka-shi, Gunma
  - Novo Nordisk Investigational Site, Chitose, Hokkaido
  - Novo Nordisk Investigational Site, Chuo-ku Tokyo
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Chūōku
  - Novo Nordisk Investigational Site, Fukuoka-shi, Fukuoka
  - Novo Nordisk Investigational Site, Higashiosaka-shi, Osaka
  - Novo Nordisk Investigational Site, Hokkaido
  - Novo Nordisk Investigational Site, Ichikawa-shi, Chiba
  - Novo Nordisk Investigational Site, Iruma-shi, Saitama
  - Novo Nordisk Investigational Site, Izumisano
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Kawagoe-shi, Saitama
  - Novo Nordisk Investigational Site, Kobe-shi, Hyogo
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Mito-shi, Ibaraki
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Neyagawa-shi, Osaka
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hygo
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hyogo
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Saga-shi,Saga
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Sappro-shi, Hokkaido
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Takatsuki-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Yokohama
  - Novo Nordisk Investigational Site, Yokohama, Kanagawa
  - Novo Nordisk Investigational Site, Yokohama-shi Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://www.novonordisk-trials.com/website/content/how-to-access-clinical-trial-datasets.aspx

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 47 sites in Japan: 47 sites screened and 45 of them randomised subjects. After screening, 635 subjects entered into the 12-week run-in period.
Pre-assignment Details: Subjects received liraglutide 0.9 mg/day (starting with 0.3 mg/day with subsequent weekly dose escalation of 0.3 mg to a maximum 0.9 mg/day) during 12 weeks run-in period. Subjects with HbA1c ≥7.0% at the end of run-in period were randomised (1:1) to two treatment arms: continuing liraglutide 0.9 mg/day or dose escalation to liraglutide 1.8 mg/day.
Groups:
- Liraglutide 1.8 mg: Subjects received liraglutide once daily subcutaneous (s.c.; under the skin) injections for 52 weeks (26-week main + 26-week extension treatment period). After the 12-week run-in period, liraglutide dose was escalated from 0.9 mg/day to 1.2 mg/day for one week, followed by a weekly dose escalation of 0.3 mg to a maximum dose of 1.8 mg/day. Subjects continued liraglutide 1.8 mg/day till week 52.
- Liraglutide 0.9 mg: Subjects received liraglutide once daily s.c. injections for 26 weeks (main treatment period). After the 12-week run-in period, subjects continued their liraglutide treatment unchanged (i.e., 0.9 mg/day) till week 26.
Period: Main Treatment Period
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Started | 233 | 233
Completed | 218 | 194
Not Completed | 15 | 39
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 7 | 17
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Unclassified | 4 | 10
Period: Extension Treatment Period
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Started | 212 (6 subjects withdrew from the trial after the main period and prior to entering the extension period) | 0 (This treatment arm is not considered for this period as the subjects were treated for 26 weeks)
Completed | 194 | 0
Not Completed | 18 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Lack of Efficacy | 4 | 0
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Unclassified | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS), which included all randomised subjects.
Groups:
- Liraglutide 1.8 mg: Subjects received liraglutide once daily s.c. injections for 52 weeks (26-week main + 26-week extension treatment period). After the 12-week run-in period, liraglutide dose was escalated from 0.9 mg/day to 1.2 mg/day for one week, followed by a weekly dose escalation of 0.3 mg to a maximum dose of 1.8 mg/day. Subjects continued liraglutide 1.8 mg/day till week 52.
- Total: Total of all reporting groups
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg | Total
Number analyzed (Participants) | 233 | 233 | 466
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.07 (10.27) | 54.96 (10.61) | 55.01 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 68 | 145
  Male | 156 | 165 | 321
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 233 | 233 | 466
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage (%) of HbA1c] | 8.14 (1.02) | 8.10 (0.87) | 8.12 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c) (Week 26)
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated after 26 weeks of treatment. The change from baseline in the response after 26 weeks of treatment is analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline response as a covariate.
Time Frame: Week 0, Week 26
Population: FAS, which included all randomised subjects. Missing values were imputed using the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%) of HbA1c
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Percentage (%) of HbA1c | -0.23 (0.06) | 0.17 (0.06)
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Liraglutide 0.9 mg; Missing data was imputed using the LOCF method. The change from baseline in the response after 26 weeks of treatment was analysed using an ANCOVA model with treatment as a fixed effect and baseline response as a covariate; Test type: Superiority — Superiority of liraglutide 1.8 mg/day vs. liraglutide 0.9 mg/day was to be considered confirmed if the 95% confidence interval for the treatment difference (liraglutide 1.8 mg/day minus liraglutide 0.9 mg/day) for change from baseline in HbA1c (% of HbA1c) was entirely below 0%, equivalent to a one-sided test with significance level of 2.5%; p < 0.0001, ANCOVA; Treatment difference = -0.40, 95% CI 2-sided [-0.55 to -0.24]

2. Secondary Outcome: Change in HbA1c (Week 52)
Description: Change from baseline (week 0) in HbA1c was evaluated after 52 weeks of treatment.
Time Frame: Week 0, Week 52
Population: FAS, which included all randomised subjects. 'Liraglutide 0.9 mg treatment arm' is not applicable for this outcome measure, as the subjects in this treatment arm received treatment for 26 weeks (main period). Missing values were imputed using the LOCF method.
Measure: Mean (Standard Deviation); unit: Percentage (%) of HbA1c
Arm/Group | Liraglutide 1.8 mg
Number analyzed (Participants) | 233
Percentage (%) of HbA1c
  Week 0: Baseline | 8.14 (1.02)
  Week 52: Change from baseline | -0.09 (1.05)

3. Secondary Outcome: Responder for HbA1c Below 7.0% (53 mmol/Mol)
Description: Reported results are number of subjects who achieved HbA1c target below 7.0% after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: FAS, which included all randomised subjects. 'Liraglutide 0.9 mg treatment arm' is not applicable for week 52, as the subjects in this treatment arm received treatment for 26 weeks (main period). Missing HbA1c values were imputed using the LOCF method.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Participants
  Week 26 | 53 | 18
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 45 |

4. Secondary Outcome: Responder for HbA1c Below or Equal to 6.5% (48 mmol/Mol)
Description: Reported results are number of subjects who achieved HbA1c target below or equal to 6.5% after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Participants
  Week 26 | 18 | 5
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 16 |

5. Secondary Outcome: Responder for HbA1c Below 7.0% Without Weight Gain
Description: Reported results are number of subjects who achieved HbA1c target below 7.0% without weight gain after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: FAS, which included all randomised subjects. 'Liraglutide 0.9 mg treatment arm' is not applicable for week 52, as the subjects in this treatment arm received treatment for 26 weeks (main period). Missing HbA1c and body weight values were imputed using the LOCF method.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Participants
  Week 26 | 36 | 13
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 35 |

6. Secondary Outcome: Responder for HbA1c Below 7.0% Without Treatment Emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Reported results are subjects with HbA1c <7.0% after 26 weeks and 52 weeks of treatment, respectively without treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes. Severe or BG confirmed symptomatic hypoglycaemia: severe as per ADA classification or BG confirmed by plasma glucose (PG) value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Severe hypoglycaemia as per ADA: episode requiring assistance of another person to actively administer carbohydrate/glucagon, or take other corrective actions. PG levels may not be available during an event, but neurological recovery following the return of PG to normal is considered sufficient evidence that the event was induced by a low PG level. Treatment emergent: episode with onset date on or after randomisation (from week (wk)0) and no later than 7 days after the last day on liraglutide (maximum till wk26+7days and wk52+7days). Hence, the following shown 'Time Frame' should be read as 'Wk26+7days and Wk52+7days'
Time Frame: Week 26 and Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Participants
  Week 26 | 53 | 18
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 45 |

7. Secondary Outcome: Change in Self-Measured Blood Glucose (SMBG) 7-point Profile: 7-point Profile (Individual Points in the Profile)
Description: Reported results are 7-point SMBG values at week 0, week 26 and week 52. The 7-point profile blood glucose levels were measured at the following time points always starting with the first:
  1. Before breakfast.
  2. 90 minutes after start of breakfast.
  3. Before lunch.
  4. 90 minutes after start of lunch.
  5. Before dinner.
  6. 90 minutes after start of dinner.
  7. At bedtime.
Time Frame: Week 0 and Week 26 and Week 52
Population: FAS, which included all randomised subjects. Number analyzed = number of subjects contributed to the analysis. 'Liraglutide 0.9 mg treatment arm' is not applicable for week 52, as the subjects in this treatment arm received treatment for 26 weeks (main period). Missing values were imputed using the LOCF method
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 0: Before breakfast: number analyzed (Participants) | 232 | 232
  Week 0: Before breakfast | 181.8 (42.8) | 177.1 (43.4)
  Week 0: 90 minutes after start of breakfast: number analyzed (Participants) | 230 | 230
  Week 0: 90 minutes after start of breakfast | 262.6 (65.0) | 266.5 (70.0)
  Week 0: Before lunch: number analyzed (Participants) | 232 | 230
  Week 0: Before lunch | 169.5 (57.7) | 177.6 (61.7)
  Week 0: 90 minutes after start of lunch: number analyzed (Participants) | 231 | 230
  Week 0: 90 minutes after start of lunch | 253.1 (64.5) | 252.2 (63.5)
  Week 0: Before dinner: number analyzed (Participants) | 231 | 230
  Week 0: Before dinner | 173.4 (59.2) | 169.7 (56.5)
  Week 0: 90 minutes after start of dinner: number analyzed (Participants) | 232 | 229
  Week 0: 90 minutes after start of dinner | 254.3 (66.2) | 249.5 (63.2)
  Week 0: At bedtime: number analyzed (Participants) | 230 | 228
  Week 0: At bedtime | 226.1 (67.4) | 217.8 (58.7)
  Week 26: Before breakfast: number analyzed (Participants) | 232 | 233
  Week 26: Before breakfast | 171.7 (39.6) | 178.2 (44.4)
  Week 26: 90 minutes after start of breakfast: number analyzed (Participants) | 232 | 233
  Week 26: 90 minutes after start of breakfast | 247.2 (64.6) | 258.2 (63.7)
  Week 26: Before lunch: number analyzed (Participants) | 231 | 232
  Week 26: Before lunch | 161.2 (51.0) | 177.0 (57.9)
  Week 26: 90 minutes after start of lunch: number analyzed (Participants) | 232 | 233
  Week 26: 90 minutes after start of lunch | 234.7 (63.3) | 255.3 (66.7)
  Week 26: Before dinner: number analyzed (Participants) | 232 | 233
  Week 26: Before dinner | 162.3 (47.5) | 168.6 (57.5)
  Week 26: 90 minutes after start of dinner: number analyzed (Participants) | 232 | 233
  Week 26: 90 minutes after start of dinner | 233.3 (60.1) | 251.5 (64.9)
  Week 26: At bedtime: number analyzed (Participants) | 231 | 232
  Week 26: At bedtime | 205.6 (58.6) | 220.5 (68.8)
  Week 52: Before breakfast: number analyzed (Participants) | 232 | 0
  Week 52: Before breakfast | 176.1 (43.2) |
  Week 52: 90 minutes after start of breakfast: number analyzed (Participants) | 229 | 0
  Week 52: 90 minutes after start of breakfast | 251.1 (69.1) |
  Week 52: Before lunch: number analyzed (Participants) | 231 | 0
  Week 52: Before lunch | 169.6 (59.7) |
  Week 52: 90 minutes after start of lunch: number analyzed (Participants) | 231 | 0
  Week 52: 90 minutes after start of lunch | 243.3 (63.9) |
  Week 52: Before dinner: number analyzed (Participants) | 232 | 0
  Week 52: Before dinner | 164.3 (50.8) |
  Week 52: 90 minutes after start of dinner: number analyzed (Participants) | 230 | 0
  Week 52: 90 minutes after start of dinner | 240.5 (65.8) |
  Week 52: At bedtime: number analyzed (Participants) | 230 | 0
  Week 52: At bedtime | 207.9 (66.7) |

8. Secondary Outcome: Change in SMBG 7-point Profile: Mean of 7-point Profile
Description: Change from baseline (week 0) in mean of the SMBG 7-point profile was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Baseline (week 0): number analyzed (Participants) | 232 | 233
  Baseline (week 0) | 217.9 (46.7) | 217.7 (46.8)
  Change from baseline: week 26: number analyzed (Participants) | 232 | 233
  Change from baseline: week 26 | -14.5 (39.0) | -0.6 (45.0)
  Change from baseline: week 52: number analyzed (Participants) | 232 | 0
  Change from baseline: week 52 | -8.9 (43.7) |

9. Secondary Outcome: Change in SMBG 7-point Profile: Mean of Postprandial Increments (From Before Meal to 90 Minutes After for Breakfast, Lunch and Dinner)
Description: Change from baseline (week 0) in mean of postprandial increments (from before meal to 90 minutes after for breakfast, lunch and dinner) of the SMBG 7-point profile was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 0: Baseline: number analyzed (Participants) | 232 | 232
  Week 0: Baseline | 81.7 (38.7) | 81.6 (38.6)
  Week 26: Change from baseline: number analyzed (Participants) | 232 | 232
  Week 26: Change from baseline | -8.4 (43.8) | -1.5 (39.5)
  Week 52: Change from baseline: number analyzed (Participants) | 232 | 0
  Week 52: Change from baseline | -6.3 (44.4) |

10. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: FAS, which included all randomised subjects. 'Liraglutide 0.9 mg treatment arm' is not applicable for week 52, as the subjects in this treatment arm received treatment for 26 weeks (main period). Missing values were imputed using the LOCF method.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 0: Baseline | 172.5 (38.7) | 172.0 (38.3)
  Week 26: Change from baseline | -8.4 (36.7) | 1.0 (33.7)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -1.2 (39.0) |

11. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Centimeter (cm)
  Week 0: Baseline | 93.68 (11.75) | 93.82 (11.50)
  Week 26: Change from baseline | -0.44 (3.04) | -0.73 (3.03)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -1.07 (3.64) |

12. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) in body weight was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Kilogram (kg)
  Week 0: Baseline | 74.67 (15.24) | 75.13 (16.46)
  Week 26: Change from baseline | -0.77 (2.01) | -0.95 (2.19)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -1.05 (2.26) |

13. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change from baseline (week 0) in BMI was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
kg/m^2
  Week 0: Baseline | 27.34 (4.80) | 27.20 (4.72)
  Week 26: Change from baseline | -0.28 (0.72) | -0.33 (0.78)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -0.39 (0.82) |

14. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic)
Description: Change from baseline (week 0) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mmHg
  Week 0: SBP, Baseline | 128.0 (13.1) | 128.8 (13.1)
  Week 26: SBP, change from baseline | -1.7 (12.8) | 0.4 (12.2)
  Week 52: SBP, change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: SBP, change from baseline | -0.9 (12.5) |
  Week 0: DBP, Baseline | 79.6 (9.1) | 80.3 (9.8)
  Week 26: DBP, change from baseline | -0.9 (8.7) | 0.1 (7.8)
  Week 52: DBP, change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: DBP, change from baseline | -0.6 (8.4) |

15. Secondary Outcome: Fasting C-peptide
Description: Fasting C-peptide was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
ng/mL
  Week 26 | 1.946 (41.9) | 1.853 (40.8)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 1.906 (42.2) |

16. Secondary Outcome: Fasting Insulin
Description: Fasting insulin was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
pmol/L
  Week 26 | 77.00 (70.9) | 70.91 (65.3)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 77.31 (68.7) |

17. Secondary Outcome: Fasting Glucagon
Description: Fasting glucagon was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
pmol/L
  Week 26 | 22.5 (30.0) | 23.4 (26.8)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 23.4 (30.2) |

18. Secondary Outcome: Proinsulin
Description: Proinsulin was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
pmol/L
  Week 26 | 15.638 (111.2) | 16.054 (101.8)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 16.217 (107.4) |

19. Secondary Outcome: Proinsulin/Insulin
Description: Proinsulin/insulin was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage (%) of proinsulin/insulin
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Percentage (%) of proinsulin/insulin
  Week 26 | 20.31 (70.7) | 22.64 (70.6)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 20.98 (72.5) |

20. Secondary Outcome: Homeostasis Model Assessment of Beta-cell Function (HOMA-B)
Description: HOMA-B was evaluated after 26 weeks and 52 weeks of treatment, respectively. HOMA-B is an index of beta-cell function and was calculated as: HOMA-B=[(20 x fasting insulin in µU/mL)/(FPG in mmol/L-3.5)].
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage (%) of beta-cell function
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Percentage (%) of beta-cell function
  Week 26 | 42.06 (73.0) | 35.54 (72.9)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 40.03 (79.5) |

21. Secondary Outcome: Homeostasis Model Assessment as an Index of Insulin Resistance (HOMA-IR)
Description: HOMA-IR was evaluated after 26 weeks and 52 weeks of treatment, respectively. HOMA-IR is an index of insulin resistance and was calculated as: HOMA-IR= fasting insulin (μU/mL) x FPG (mmol/L)/22.5.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: HOMA-IR score
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
HOMA-IR score
  Week 26 | 4.388 (81.9) | 4.262 (73.5)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 4.567 (77.5) |

22. Secondary Outcome: Total Cholesterol
Description: Total cholesterol was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 26 | 191.2 (17.6) | 194.5 (16.1)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 190.6 (16.3) |

23. Secondary Outcome: Low Density Lipoprotein (LDL) Cholesterol
Description: LDL was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 26 | 103.4 (31.6) | 107.1 (27.8)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 104.5 (26.2) |

24. Secondary Outcome: High Density Lipoprotein (HDL) Cholesterol
Description: HDL was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 26 | 52.7 (25.6) | 52.9 (26.3)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 53.3 (24.7) |

25. Secondary Outcome: Very Low Density Lipoprotein (VLDL) Cholesterol
Description: VLDL was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 26 | 26.8 (56.7) | 27.8 (49.4)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 25.9 (55.2) |

26. Secondary Outcome: Triglycerides
Description: Triglycerides were evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 26 | 135.4 (60.1) | 142.3 (54.9)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 130.4 (57.0) |

27. Secondary Outcome: Free Fatty Acids
Description: Free fatty acids were evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 26 and Week 52
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 26 | 12.56 (47.4) | 12.99 (43.9)
  Week 52: number analyzed (Participants) | 233 | 0
  Week 52 | 12.19 (44.3) |

28. Secondary Outcome: Number of Treatment Emergent Adverse Events
Description: Treatment emergent adverse events (TEAEs) were evaluated during the 26-week and 52-week treatment period, respectively. TEAE for weeks 0-26: Event that has onset date on or after randomisation (from week 0) and no later than seven days after the last day on liraglutide (maximum till week 26 + 7 days). TEAE for weeks 0-52: Event that has onset date on or after randomisation (from week 0) and no later than seven days after the last day on liraglutide (maximum till week 52 + 7 days). Hence, the following shown 'Time Frame' should be read as 'Weeks 0-26 + 7 days and Weeks 0-52 + 7 days'.
Time Frame: Weeks 0-26 and Weeks 0-52
Population: Safety analysis set, which included all subjects receiving at least one dose of liraglutide. 'Liraglutide 0.9 mg treatment arm' is not applicable for weeks 0-52, as the subjects in this treatment arm received treatment for 26 weeks (main period).
Measure: Number; unit: Events
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Events
  Weeks 0-26 | 365 | 266
  Weeks 0-52: number analyzed (Participants) | 233 | 0
  Weeks 0-52 | 588 |

29. Secondary Outcome: Number of Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were evaluated during the 26-week and 52-week treatment period, respectively. Severe or BG confirmed symptomatic hypoglycaemia (hypo):An episode that was severe according to the ADA classification or BG confirmed by a PG value <3.1 mmol/L with symptoms consistent with hypo. ADA definition of severe hypo:episode requiring assistance of another person to actively administer carbohydrate/glucagon, or take other corrective actions. PG levels may not be available during an event, but neurological recovery following the return of PG to normal is considered sufficient evidence that the event was induced by a low PG level. Treatment emergent: episode with onset date on or after randomisation (from week (wk) 0) and no later than 7 days after the last day on liraglutide (maximum till wk 26 and wk 52, respectively + 7 days). Hence, the following shown 'Time Frame' should be read as 'wk 0-26+7 days and wk 0-52+7 days'.
Time Frame: Weeks 0-26 and Weeks 0-52
Population: as for outcome 28
Measure: Number; unit: Episodes
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Episodes
  Weeks 0-26 | 0 | 0
  Weeks 0-52: number analyzed (Participants) | 233 | 0
  Weeks 0-52 | 0 |

30. Secondary Outcome: Number of Treatment Emergent Nocturnal Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent nocturnal severe or BG confirmed symptomatic hypoglycaemic episodes were evaluated during the26-week and 52-week treatment period, respectively. Nocturnal hypoglycaemic episodes: Those occurring between 00:01 and 05:59 hours, both inclusive. Severe or BG confirmed symptomatic hypoglycaemia: episode that was severe according to the ADA classification or BG confirmed by a PG value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Treatment emergent: episode with onset date on or after randomisation (from week 0) and no later than 7 days after the last day on liraglutide (maximum till week 26 and week 52, respectively + 7 days). Hence, the following shown 'Time Frame' should be read as 'Week 0-26 + 7 days and Week 0-52 + 7 days'.
Time Frame: Weeks 0-26 and Weeks 0-52
Population: Safety analysis set, which included all subjects receiving at least one dose of liraglutide. 'Liraglutide 0.9 mg treatment arm' is not applicable for week 52, as the subjects in this treatment arm received treatment for 26 weeks (main period).
Measure: Number; unit: Episodes
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Episodes
  Weeks 0-26 | 0 | 0
  Weeks 0-52: number analyzed (Participants) | 233 | 0
  Weeks 0-52 | 0 |

31. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to ADA Definition
Description: American Diabetes Association (ADA) classification of hypoglycaemia:
  1. Severe: Requiring assistance of another person to actively administer carbohydrate/glucagon/take other corrective actions. PG levels may not be available during an event, but neurological recovery following return of PG to normal is considered sufficient evidence that event was induced by a low PG level.
  2. Documented symptomatic: PG level ≤3.9 mmol/L with symptoms.
  3. Asymptomatic: PG level ≤3.9 mmol/L without symptoms.
  4. Probable symptomatic: No measurement with symptoms.
  5. Pseudo: PG level >3.9 mmol/L with symptoms. Treatment emergent hypoglycaemic episode: episode with onset date on or after randomisation (from week 0) and no later than 7 days after the last day on liraglutide (maximum till week 26 and week 52, respectively + 7 days). Hence, the following shown 'Time Frame' should be read as 'Week 0-26 + 7 days and Week 0-52 + 7 days'.
Time Frame: Weeks 0-26 and Weeks 0-52
Population: as for outcome 30
Measure: Number; unit: Episodes
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Episodes
  Weeks 0-26: Severe hypoglycaemia | 0 | 0
  Weeks 0-26: Documented symptomatic hypoglycaemia | 0 | 0
  Weeks 0-26: Asymptomatic hypoglycaemia | 2 | 1
  Weeks 0-26: Probable symptomatic hypoglycaemia | 3 | 1
  Weeks 0-26: Pseudo-hypoglycaemia | 2 | 1
  Weeks 0-52: Severe hypoglycaemia: number analyzed (Participants) | 233 | 0
  Weeks 0-52: Severe hypoglycaemia | 0 |
  Weeks 0-52: Documented symptomatic hypoglycaemia: number analyzed (Participants) | 233 | 0
  Weeks 0-52: Documented symptomatic hypoglycaemia | 0 |
  Weeks 0-52: Asymptomatic hypoglycaemia: number analyzed (Participants) | 233 | 0
  Weeks 0-52: Asymptomatic hypoglycaemia | 3 |
  Weeks 0-52: Probable symptomatic hypoglycaemia: number analyzed (Participants) | 233 | 0
  Weeks 0-52: Probable symptomatic hypoglycaemia | 4 |
  Weeks 0-52: Pseudo-hypoglycaemia: number analyzed (Participants) | 233 | 0
  Weeks 0-52: Pseudo-hypoglycaemia | 2 |

32. Secondary Outcome: Change in Pulse
Description: Change from baseline (week 0) in pulse was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: Safety analysis set, which included all subjects receiving at least one dose of liraglutide. 'Liraglutide 0.9 mg treatment arm' is not applicable for week 52, as the subjects in this treatment arm received treatment for 26 weeks (main period). Missing values were imputed using the LOCF method.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Beats/minute
  Week 0: Baseline | 80.2 (9.8) | 80.8 (10.4)
  Week 26: Change from baseline | 0.8 (7.8) | 0.2 (7.9)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.2 (8.1) |

33. Secondary Outcome: Change in Physical Examination
Description: Reported results are physical examination outcomes at week (wk) 0, wk 26 and wk 52. Physical examination consisted of the following listed examinations and the outcome of each examination was evaluated as: 1) normal, 2) abnormal, not clinically significant (NCS) or 3) abnormal, clinically significant (CS).
  1. Cardiovascular system
  2. Central and peripheral nervous system (PNS)
  3. Gastrointestinal (GI) system including mouth
  4. General appearance
  5. Head, ears, eyes, nose, throat, neck
  6. Lymph node palpation
  7. Musculoskeletal system
  8. Respiratory system
  9. Skin
  10. Thyroid gland
Time Frame: Week 0 and Week 26 and Week 52
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Participants
  Cardiovascular system: Wk 0: Normal | 229 | 230
  Cardiovascular system: Wk 0: Abnormal, NCS | 3 | 0
  Cardiovascular system: Wk 0: Abnormal, CS | 1 | 3
  Cardiovascular system: Wk 26: Normal | 230 | 229
  Cardiovascular system: Wk 26: Abnormal, NCS | 2 | 0
  Cardiovascular system: Week 26: Abnormal, CS | 1 | 4
  Cardiovascular system: Wk 52: Normal: number analyzed (Participants) | 233 | 0
  Cardiovascular system: Wk 52: Normal | 227 |
  Cardiovascular system: Wk 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Cardiovascular system: Wk 52: Abnormal, NCS | 4 |
  Cardiovascular system: Wk 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  Cardiovascular system: Wk 52: Abnormal, CS | 2 |
  Central and PNS: Wk 0: Normal | 232 | 229
  Central and PNS: Wk 0: Abnormal, NCS | 0 | 1
  Central and PNS: Wk 0: Abnormal, CS | 1 | 3
  Central and PNS: Wk 26: Normal | 231 | 229
  Central and PNS: Wk 26: Abnormal, NCS | 0 | 1
  Central and PNS: Wk 26: Abnormal, CS | 2 | 3
  Central and PNS: Wk 52: Normal: number analyzed (Participants) | 233 | 0
  Central and PNS: Wk 52: Normal | 232 |
  Central and PNS: Wk 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Central and PNS: Wk 52: Abnormal, NCS | 0 |
  Central and PNS: Wk 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  Central and PNS: Wk 52: Abnormal, CS | 1 |
  GI system including mouth: Wk 0: Normal | 227 | 226
  GI system including mouth: Wk 0: Abnormal, NCS | 0 | 4
  GI system including mouth: Wk 0: Abnormal, CS | 6 | 3
  GI system including mouth: Wk 26: Normal | 227 | 226
  GI system including mouth: Wk 26: Abnormal, NCS | 0 | 3
  GI system including mouth: Wk 26: Abnormal, CS | 6 | 4
  GI system including mouth: Wk 52: Normal: number analyzed (Participants) | 233 | 0
  GI system including mouth: Wk 52: Normal | 226 |
  GI system including mouth: Wk 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  GI system including mouth: Wk 52: Abnormal, NCS | 2 |
  GI system including mouth: Wk 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  GI system including mouth: Wk 52: Abnormal, CS | 5 |
  General appearance: Wk 0: Normal | 229 | 232
  General appearance: Wk 0: Abnormal, NCS | 4 | 1
  General appearance: Wk 0: Abnormal, CS | 0 | 0
  General appearance: Wk 26: Normal | 229 | 233
  General appearance: Wk 26: Abnormal, NCS | 4 | 0
  General appearance: Wk 26: Abnormal, CS | 0 | 0
  General appearance: Wk 52: Normal: number analyzed (Participants) | 233 | 0
  General appearance: Wk 52: Normal | 229 |
  General appearance: Wk 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  General appearance: Wk 52: Abnormal, NCS | 4 |
  General appearance: Wk 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  General appearance: Wk 52: Abnormal, CS | 0 |
  Head,ears,eyes,nose,throat,neck: Wk0:Normal | 225 | 226
  Head,ears,eyes,nose,throat,neck: Wk0:Abnormal,NCS | 3 | 2
  Head,ears,eyes,nose,throat,neck: Wk0:Abnormal,CS | 5 | 5
  Head,ears,eyes,nose,throat,neck: Wk26:Normal | 225 | 228
  Head,ears,eyes,nose,throat,neck: Wk26:Abnormal,NCS | 4 | 1
  Head,ears,eyes,nose,throat,neck: Wk26:Abnormal,CS | 4 | 4
  Head,ears,eyes,nose,throat,neck: Wk52:Normal: number analyzed (Participants) | 233 | 0
  Head,ears,eyes,nose,throat,neck: Wk52:Normal | 223 |
  Head,ears,eyes,nose,throat,neck: Wk52:Abnormal,NCS: number analyzed (Participants) | 233 | 0
  Head,ears,eyes,nose,throat,neck: Wk52:Abnormal,NCS | 5 |
  Head,ears,eyes,nose,throat,neck: Wk52:Abnormal,CS: number analyzed (Participants) | 233 | 0
  Head,ears,eyes,nose,throat,neck: Wk52:Abnormal,CS | 5 |
  Lymph node palpation: Wk 0: Normal | 233 | 233
  Lymph node palpation: Wk 0: Abnormal, NCS | 0 | 0
  Lymph node palpation: Wk 0: Abnormal, CS | 0 | 0
  Lymph node palpation: Wk 26: Normal | 233 | 233
  Lymph node palpation: Wk 26: Abnormal, NCS | 0 | 0
  Lymph node palpation: Wk 26: Abnormal, CS | 0 | 0
  Lymph node palpation: Wk 52: Normal: number analyzed (Participants) | 233 | 0
  Lymph node palpation: Wk 52: Normal | 233 |
  Lymph node palpation: Wk 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Lymph node palpation: Wk 52: Abnormal, NCS | 0 |
  Lymph node palpation: Wk 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  Lymph node palpation: Wk 52: Abnormal, CS | 0 |
  Musculoskeletal system: Wk 0: Normal | 226 | 231
  Musculoskeletal system: Wk 0: Abnormal, NCS | 4 | 0
  Musculoskeletal system: Wk 0: Abnormal, CS | 3 | 2
  Musculoskeletal system: Wk 26: Normal | 224 | 230
  Musculoskeletal system: Wk 26: Abnormal, NCS | 5 | 0
  Musculoskeletal system: Wk 26: Abnormal, CS | 4 | 3
  Musculoskeletal system: Wk 52: Normal: number analyzed (Participants) | 233 | 0
  Musculoskeletal system: Wk 52: Normal | 224 |
  Musculoskeletal system: Wk 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Musculoskeletal system: Wk 52: Abnormal, NCS | 5 |
  Musculoskeletal system: Wk 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  Musculoskeletal system: Wk 52: Abnormal, CS | 4 |
  Respiratory system: Wk 0: Normal | 233 | 232
  Respiratory system: Wk 0: Abnormal, NCS | 0 | 1
  Respiratory system: Wk 0: Abnormal, CS | 0 | 0
  Respiratory system: Wk 26: Normal | 232 | 232
  Respiratory system: Wk 26: Abnormal, NCS | 0 | 1
  Respiratory system: Wk 26: Abnormal, CS | 1 | 0
  Respiratory system: Wk 52: Normal: number analyzed (Participants) | 233 | 0
  Respiratory system: Wk 52: Normal | 232 |
  Respiratory system: Wk 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Respiratory system: Wk 52: Abnormal, NCS | 0 |
  Respiratory system: Wk 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  Respiratory system: Wk 52: Abnormal, CS | 1 |
  Skin: Wk 0: Normal | 225 | 223
  Skin: Wk 0: Abnormal, NCS | 4 | 3
  Skin: Wk 0: Abnormal, CS | 4 | 7
  Skin: Wk 26: Normal | 218 | 222
  Skin: Wk 26: Abnormal, NCS | 4 | 4
  Skin: Wk 26: Abnormal, CS | 11 | 7
  Skin: Wk 52: Normal: number analyzed (Participants) | 233 | 0
  Skin: Wk 52: Normal | 224 |
  Skin: Wk 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Skin: Wk 52: Abnormal, NCS | 4 |
  Skin: Wk 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  Skin: Wk 52: Abnormal, CS | 5 |
  Thyroid gland: Wk 0: Normal | 232 | 232
  Thyroid gland: Wk 0: Abnormal, NCS | 0 | 0
  Thyroid gland: Wk 0: Abnormal, CS | 1 | 1
  Thyroid gland: Wk 26: Normal | 232 | 232
  Thyroid gland: Wk 26: Abnormal, NCS | 0 | 0
  Thyroid gland: Wk 26: Abnormal, CS | 1 | 1
  Thyroid gland: Wk 52: Normal: number analyzed (Participants) | 233 | 0
  Thyroid gland: Wk 52: Normal | 232 |
  Thyroid gland: Wk 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Thyroid gland: Wk 52: Abnormal, NCS | 0 |
  Thyroid gland: Wk 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  Thyroid gland: Wk 52: Abnormal, CS | 1 |

34. Secondary Outcome: Change in Eye Examination
Description: Reported results are eye examination (ophthalmoscopy) outcomes at week 0, week 26 and week 52. Ophthalmoscopy outcomes for both left and right eye were evaluated as: 1) normal, 2) abnormal, NCS or 3) abnormal, CS.
Time Frame: Week 0 and Week 26 and Week 52
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Participants
  Week 0: Left eye - Normal | 183 | 176
  Week 0: Left eye - Abnormal, NCS | 15 | 13
  Week 0: Left eye - Abnormal, CS | 35 | 44
  Week 26: Left eye - Normal | 178 | 178
  Week 26: Left eye - Abnormal, NCS | 18 | 15
  Week 26: Left eye - Abnormal, CS | 37 | 40
  Week 52: Left eye - Normal: number analyzed (Participants) | 233 | 0
  Week 52: Left eye - Normal | 181 |
  Week 52: Left eye - Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Week 52: Left eye - Abnormal, NCS | 16 |
  Week 52: Left eye - Abnormal, CS: number analyzed (Participants) | 233 | 0
  Week 52: Left eye - Abnormal, CS | 36 |
  Week 0: Right eye - Normal | 183 | 180
  Week 0: Right eye - Abnormal, NCS | 14 | 11
  Week 0: Right eye - Abnormal, CS | 36 | 42
  Week 26: Right eye - Normal | 176 | 180
  Week 26: Right eye - Abnormal, NCS | 19 | 14
  Week 26: Right eye - Abnormal, CS | 38 | 39
  Week 52: Right eye - Normal: number analyzed (Participants) | 233 | 0
  Week 52: Right eye - Normal | 177 |
  Week 52: Right eye - Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Week 52: Right eye - Abnormal, NCS | 18 |
  Week 52: Right eye - Abnormal, CS: number analyzed (Participants) | 233 | 0
  Week 52: Right eye - Abnormal, CS | 38 |

35. Secondary Outcome: Change in Electrocardiogram (ECG)
Description: Reported results are ECG outcomes at week 0, week 26 and week 52. ECG outcomes were evaluated as: 1) normal, 2) abnormal, NCS or 3) abnormal, CS.
Time Frame: Week 0 and Week 26 and Week 52
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Participants
  Week 0: Normal | 202 | 196
  Week 0: Abnormal, NCS | 31 | 35
  Week 0: Abnormal, CS | 0 | 2
  Week 26: Normal | 205 | 204
  Week 26: Abnormal, NCS | 26 | 26
  Week 26: Abnormal, CS | 2 | 3
  Week 52: Normal: number analyzed (Participants) | 233 | 0
  Week 52: Normal | 203 |
  Week 52: Abnormal, NCS: number analyzed (Participants) | 233 | 0
  Week 52: Abnormal, NCS | 28 |
  Week 52: Abnormal, CS: number analyzed (Participants) | 233 | 0
  Week 52: Abnormal, CS | 2 |

36. Secondary Outcome: Change in Biochemistry: Creatinine
Description: Change from baseline (week 0) in creatinine was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 0: Baseline | 0.802 (0.144) | 0.822 (0.164)
  Week 26: Change from baseline | 0.018 (0.070) | 0.011 (0.080)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.025 (0.078) |

37. Secondary Outcome: Change in Biochemistry: eGFR
Description: Change from baseline (week 0) in estimated glomerular filtration rate (eGFR) was evaluated after 26 weeks and 52 weeks of treatment, respectively. eGFR was evaluated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula, mL/min/1.73m^2.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mL/min/1.73m^2
  Week 0: Baseline | 78.6 (9.5) | 77.6 (10.7)
  Week 26: Change from baseline | -1.5 (5.0) | -1.0 (5.8)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -2.3 (5.6) |

38. Secondary Outcome: Change in Biochemistry: Alanine Aminotransferase
Description: Change from baseline (week 0) in alanine aminotransferase was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
U/L
  Week 0: Baseline | 32.7 (19.5) | 34.2 (21.8)
  Week 26: Change from baseline | -0.4 (12.0) | -2.2 (13.9)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -2.4 (11.9) |

39. Secondary Outcome: Change in Biochemistry: Aspartate Aminotransferase
Description: Change from baseline (week 0) in aspartate aminotransferase was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
U/L
  Week 0: Baseline | 26.5 (12.8) | 26.9 (13.9)
  Week 26: Change from baseline | 0.2 (9.9) | -1.0 (8.6)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -1.2 (8.9) |

40. Secondary Outcome: Change in Biochemistry: Alkaline Phosphatase
Description: Change from baseline (week 0) in alkaline phosphatase was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
U/L
  Week 0: Baseline | 72.5 (20.6) | 74.1 (22.1)
  Week 26: Change from baseline | 0.6 (9.8) | 2.0 (12.4)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 2.1 (11.1) |

41. Secondary Outcome: Change in Biochemistry: Sodium
Description: Change from baseline (week 0) in sodium was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mmol/L
  Week 0: Baseline | 140.2 (1.9) | 140.2 (1.9)
  Week 26: Change from baseline | 0.1 (1.8) | 0.2 (2.0)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.3 (1.8) |

42. Secondary Outcome: Change in Biochemistry: Potassium
Description: Change from baseline (week 0) in potassium was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mmol/L
  Week 0: Baseline | 4.40 (0.34) | 4.38 (0.34)
  Week 26: Change from baseline | -0.01 (0.32) | -0.02 (0.29)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.00 (0.31) |

43. Secondary Outcome: Change in Biochemistry: Albumin
Description: Change from baseline (week 0) in albumin was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
g/L
  Week 0: Baseline | 44.7 (2.5) | 45.1 (2.2)
  Week 26: Change from baseline | -0.2 (2.1) | -0.2 (1.9)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -0.2 (2.2) |

44. Secondary Outcome: Change in Biochemistry: Total Bilirubin
Description: Change from baseline (week 0) in total bilirubin was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 0: Baseline | 0.52 (0.29) | 0.53 (0.25)
  Week 26: Change from baseline | 0.04 (0.25) | 0.04 (0.24)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.06 (0.23) |

45. Secondary Outcome: Change in Biochemistry: Urea
Description: Change from baseline (week 0) in urea was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 0: Baseline | 13.5 (3.2) | 14.0 (3.7)
  Week 26: Change from baseline | 0.3 (3.0) | -0.0 (3.3)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.7 (2.8) |

46. Secondary Outcome: Change in Biochemistry: Creatine Kinase
Description: Change from baseline (week 0) in creatine kinase was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
U/L
  Week 0: Baseline | 117.3 (61.8) | 129.3 (100.3)
  Week 26: Change from baseline | 5.2 (50.9) | -5.2 (96.3)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 7.5 (54.8) |

47. Secondary Outcome: Change in Biochemistry: Calcium
Description: Change from baseline (week 0) in calcium was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 0: Baseline | 9.66 (0.41) | 9.66 (0.37)
  Week 26: Change from baseline | -0.01 (0.41) | 0.01 (0.39)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.01 (0.41) |

48. Secondary Outcome: Change in Biochemistry: Albumin Corrected Calcium
Description: Change from baseline (week 0) in albumin corrected calcium was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
mg/dL
  Week 0: Baseline | 9.28 (0.35) | 9.26 (0.32)
  Week 26: Change from baseline | 0.00 (0.37) | 0.02 (0.35)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.02 (0.36) |

49. Secondary Outcome: Change in Biochemistry: Amylase
Description: Change from baseline (week 0) in amylase was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
U/L
  Week 0: Baseline | 62.3 (23.1) | 61.1 (22.5)
  Week 26: Change from baseline | -0.9 (12.5) | -2.3 (13.3)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -0.7 (12.1) |

50. Secondary Outcome: Change in Biochemistry: Lipase
Description: Change from baseline (week 0) in lipase was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
U/L
  Week 0: Baseline | 55.4 (26.1) | 57.3 (28.7)
  Week 26: Change from baseline | -1.4 (23.4) | -3.3 (26.7)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -1.0 (22.0) |

51. Secondary Outcome: Change in Haematology: Haemoglobin
Description: Change from baseline (week 0) in haemoglobin was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
g/dL
  Week 0: Baseline | 14.65 (1.26) | 14.56 (1.35)
  Week 26: Change from baseline | -0.00 (0.67) | 0.04 (0.57)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -0.00 (0.76) |

52. Secondary Outcome: Change in Haematology: Haematocrit
Description: Change from baseline (week 0) in haematocrit was evaluated after 26 weeks and 52 weeks of treatment, respectively. Haematocrit is the ratio of the volume of red blood cells to the total volume of blood.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: % of red blood cell
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
% of red blood cell
  Week 0: Baseline | 44.86 (3.79) | 44.65 (4.03)
  Week 26: Change from baseline | -0.22 (2.26) | -0.06 (1.90)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -0.49 (2.39) |

53. Secondary Outcome: Change in Haematology: Thrombocytes
Description: Change from baseline (week 0) in thrombocytes (platelets) was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26 and Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
10^9 cells/L
  Week 0: Baseline | 229.1 (47.4) | 231.0 (57.6)
  Week 26: Change from baseline | 0.8 (27.4) | -1.5 (24.2)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 3.4 (24.9) |

54. Secondary Outcome: Change in Haematology: Erythrocytes
Description: Change from baseline (week 0) in erythrocytes was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26 and Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
10^12 cells/L
  Week 0: Baseline | 4.87 (0.41) | 4.89 (0.43)
  Week 26: Change from baseline | -0.02 (0.24) | -0.00 (0.20)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -0.04 (0.25) |

55. Secondary Outcome: Change in Haematology: Leukocytes
Description: Change from baseline (week 0) in leukocytes was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26 and Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
10^9 cells/L
  Week 0: Baseline | 6.55 (1.71) | 6.53 (1.58)
  Week 26: Change from baseline | 0.09 (1.15) | -0.08 (1.09)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.09 (1.44) |

56. Secondary Outcome: Change in Haematology: Eosinophils
Description: Change from baseline (week 0) in eosinophils was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26 and Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
10^9 cells/L
  Week 0: Baseline | 0.182 (0.143) | 0.167 (0.158)
  Week 26: Change from baseline | 0.001 (0.118) | -0.016 (0.104)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | -0.008 (0.108) |

57. Secondary Outcome: Change in Haematology: Neutrophils
Description: Change from baseline (week 0) in neutrophils was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26 and Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
10^9 cells/L
  Week 0: Baseline | 3.967 (1.337) | 3.975 (1.236)
  Week 26: Change from baseline | 0.054 (1.029) | -0.088 (0.941)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.062 (1.239) |

58. Secondary Outcome: Change in Haematology: Basophils
Description: Change from baseline (week 0) in basophils was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26 and Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
10^9 cells/L
  Week 0: Baseline | 0.024 (0.013) | 0.026 (0.013)
  Week 26: Change from baseline | 0.004 (0.017) | 0.000 (0.016)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.000 (0.016) |

59. Secondary Outcome: Change in Haematology: Monocytes
Description: Change from baseline (week 0) in monocytes was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26 and Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
10^9 cells/L
  Week 0: Baseline | 0.341 (0.133) | 0.326 (0.120)
  Week 26: Change from baseline | 0.001 (0.101) | -0.000 (0.104)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.019 (0.153) |

60. Secondary Outcome: Change in Haematology: Lymphocytes
Description: Change from baseline (week 0) in lymphocytes was evaluated after 26 weeks and 52 weeks of treatment, respectively.
Time Frame: Week 0, Week 26 and Week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
10^9 cells/L
  Week 0: Baseline | 2.034 (0.561) | 2.037 (0.583)
  Week 26: Change from baseline | 0.032 (0.364) | 0.022 (0.389)
  Week 52: Change from baseline: number analyzed (Participants) | 233 | 0
  Week 52: Change from baseline | 0.014 (0.347) |

61. Secondary Outcome: Change in Calcitonin
Description: Reported results are number of subjects with low, normal or high calcitonin values at week 0, week 26 and week 52. Number of subjects analyzed = number of subjects contributed to the analysis for individual time point. Calcitonin values were categorised as low, normal or high.
Time Frame: Week 0 and Week 26 and Week 52
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
Number analyzed (Participants) | 233 | 233
Participants
  Week 0: Low: number analyzed (Participants) | 233 | 232
  Week 0: Low | 0 | 0
  Week 0: Normal: number analyzed (Participants) | 233 | 232
  Week 0: Normal | 229 | 229
  Week 0: High: number analyzed (Participants) | 233 | 232
  Week 0: High | 4 | 3
  Week 26: Low | 0 | 0
  Week 26: Normal | 228 | 231
  Week 26: High | 5 | 2
  Week 52: Low: number analyzed (Participants) | 233 | 0
  Week 52: Low | 0 |
  Week 52: Normal: number analyzed (Participants) | 233 | 0
  Week 52: Normal | 230 |
  Week 52: High: number analyzed (Participants) | 233 | 0
  Week 52: High | 3 |

ADVERSE EVENTS:
Time Frame: Liraglutide 1.8 mg treatment arm: Week 0 to week 52 (treatment period) + 7 days (follow-up period). Liraglutide 0.9 mg treatment arm: Week 0 to week 26 (treatment period) + 7 days (follow-up period).
Description: All presented adverse events are treatment emergent (i.e., TEAEs). A TEAE was defined as an event that has onset date on or after randomisation (from week 0) and no later than seven days after the last day on liraglutide (maximum till week 26 and week 52, respectively + 7 days). Results are based on the safety analysis set, which included all subjects receiving at least one dose of liraglutide.
Arm/Group | Liraglutide 1.8 mg | Liraglutide 0.9 mg
All-Cause Mortality (participants affected / at risk) | 0/233 | 0/233
Serious Adverse Events (participants affected / at risk) | 8/233 | 3/233
Other Adverse Events (participants affected / at risk) | 99/233 | 65/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 1.8 mg (N=233) | Liraglutide 0.9 mg (N=233)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 1.8 mg (N=233) | Liraglutide 0.9 mg (N=233)
Constipation (Gastrointestinal disorders) | 17 (19) | 5 (5)
Diabetic retinopathy (Eye disorders) | 23 (24) | 17 (17)
Viral upper respiratory tract infection (Infections and infestations) | 66 (94) | 44 (52)
Lipase increased (Investigations) | 13 (13) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT02505334/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT02505334/SAP_001.pdf